CLINICAL TRIAL: NCT05524142
Title: Association Between ALDH2 Gene Polymorphism and Atrial Fibrillation
Acronym: AAAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0404
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ALDH2
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atrial fibrillation: Patients with atrial fibrillation underwent radiofrequency ablation.
- Control: Patients underwent electrophysiological examination alone and were confirmed no arrhythmia.

SUMMARY:
This study is a case-control study. In this study, 2ml of vein blood samples were collected from patients with atrial fibrillation undergoing radiofrequency ablation and those in the control group who underwent electrophysiological examination alone and confirmed no arrhythmia. The purpose of this study is to identify the relationship between the aldehyde dehydrogenase 2 (ALDH2) gene polymorphism and susceptibility to atrial fibrillation, and to explore the relationship between the genotype of ALDH2 SNP and the prognosis of patients with atrial fibrillation undergoing radiofrequency ablation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;

  * Age 18-85 years old, gender is not limited; ③ Case group: patients with clinical diagnosis of atrial fibrillation who underwent radiofrequency ablation; control group: patients with no arrhythmia confirmed by electrophysiological examination; ④ Able to communicate well with investigators and comply with the entire trial requirements.

Exclusion Criteria:

* Those who cannot understand or refuse to sign the informed consent or follow-up; ②Pregnant women, mentally retarded, mental/cognitive insufficiency and other possible vulnerable groups

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients diagnosed with atrial fibrillation in the Second Affiliated Hospital of Zhejiang University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation recurrence | 3 months
  atrial fibrillation recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jin J, Qian N, Gao Y, Liu J, Chen D, Wang B, Luo M, Zhang Y, Ye J, Jiang R, Wang L, Jiang J, Wang Y. Diabetes and ALDH2 Gene Polymorphism on Post-Ablation Atrial Fibrillation Recurrence. JACC Asia. 2025 Nov 12:S2772-3747(25)00638-6. doi: 10.1016/j.jacasi.2025.10.021. Online ahead of print. PMID 41342828